CLINICAL TRIAL: NCT04199078
Title: Ensayo clínico Aleatorizado, Abierto, Paralelo, Controlado, multicéntrico, Para Explorar la Eficacia Del Gel Vaginal Papilocare® en la reparación de la Mucosa Cervical Con Lesiones Causadas Por Virus Papiloma Humano de Alto Riesgo
Brief Title: Clinical Trial to Explore Papilocare Gel Efficacy to Repair of the Cervico-vaginal Mucosa With HPV High Risk Lesions.
Acronym: PALOMA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procare Health Iberia S.L. (Industry)
Collaborators: Adknoma Health Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PALOMA II
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Human Papilloma Virus; Human Papilloma Virus Infection; Cervix Lesion
Keywords: HPV
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A - papilocare alternative days treatment (Experimental): Arm A: scheme A (21 days / 1 cannula per day + 7 days rest) x 1 month + alternate days up to 6 months (except for menstruation days)
  Interventions: Device: Papilocare vaginal gel
- B - papilocare semiintensive treatment (Experimental): Arm B: scheme B (21 days / 1 cannula per day + 7 days rest) x 3 months + alternate days up to 6 months (except menstruation days)
  Interventions: Device: Papilocare vaginal gel
- C - papilocare intensive treatment (Experimental): Arm C: scheme C (21 days / 1 cannula per day + 7 days rest) x 6 months
  Interventions: Device: Papilocare vaginal gel
- D - standard of care (No Intervention): Arm D: usual clinical practice - no treatment

INTERVENTIONS:
Device: Papilocare vaginal gel — Papilocare is a gel vaginally administered by a singledose cannula. Vaginal gel formulation is effective as a local treatment with controlled systemic absorption and rapid and efficient distribution
  Arms: A - papilocare alternative days treatment; B - papilocare semiintensive treatment; C - papilocare intensive treatment

SUMMARY:
Phase II, exploratory, randomized, open, controlled and parallel groups clinical trial to evaluate the effectiveness of exploratory gel Papilocare in the repair of the cervico-vaginal mucosa with lesions caused by HPV-HR. All the patients included in the study will be randomized (1:1:1:1) in 4 arms.

DETAILED DESCRIPTION:
Phase II, exploratory, randomized, open, controlled and parallel groups clinical trial to evaluate the effectiveness of exploratory gel Papilocare in the repair of the cervico-vaginal mucosa with lesions caused by HPV-HR. All the patients included in the study will be randomized (1:1:1:1) to Arm A (Papilocare schedule A), Arm B (Papilocare schedule B) and Arm C (Papilocare schedule C) Arm D (usual clinical practice-without treatment-).

Selection period of 1 month, followed by randomization and 6 months of treatment followed by a period of another 6 months without treatment.

Patients will visit the site into a total of 5 visits throughout the study. Total study duration: 13 months.

ELIGIBILITY:
Inclusion Criteria:

1. Woman between the ages of 30 and 65 (both inclusive).
2. Able to read and understand the Patient Information Sheet and the Informed Consent form.
3. Acceptance in the participation of the essay and signature of the Informed Consent form.
4. ASC-US or LSIL or AG-US cytological result (maximum 3 months prior to inclusion) with concordant colposcopic image (performed at the screening visit).
5. High risk HPV positive by PCR performed at screening visit.
6. Is able, at the discretion of the researcher, to comply with the requirements of the trial and without hindrance to follow the instructions and assessments throughout it.

Exclusion Criteria:

1. Clinically relevant immune system alterations, or any other autoimmune disease or in treatment with immunosuppressants.
2. Non-diagnosed abnormal genital hemorrhage (during the 6 months prior to the screening visit).
3. To had been vaccinated against HPV.
4. Other symptomatic vulvovaginal infections.
5. Surgical cervical excision in the last year or total hysterectomy.
6. Previous history of gynecological cancer.
7. Participation in any other clinical trial at present or in the 4 weeks prior to the inclusion of the trial.
8. Any planned surgery that prevents the correct compliance with the guidelines.
9. Use of vaginal contraceptives or other vaginal hormonal treatments.
10. Contraindications for the use of Papilocare® gel or known allergies to any of its components.
11. Women of childbearing age who do not use effective contraceptive methods, pregnant women, with suspicion of pregnancy or woman who are breastfeeding.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the repairment of the cervico-vaginal mucosa with concordant colposcopic image | 6 months
  Evaluate the repairment of the cervico-vaginal mucosa in positive high risk HPV women with a cytological result of squamous atypia of undetermined significance (ASC-US) or low-grade squamous lesion (LSIL) or glandular atypia of undetermined significance (AG-US), with concordant colposcopic image, 6 months after the start of treatment.

SECONDARY OUTCOMES:
Evaluate the repairment of the cervico-vaginal mucosa with concordant colposcopic image | 3 and 12 months
  Evaluate the repairment of the cervico-vaginal mucosa in positive high risk HPV women with a cytological result of squamous atypia of undetermined significance (ASC-US) or low-grade squamous lesion (LSIL) or glandular atypia of undetermined significance (AG-US), with concordant colposcopic image at 3 and 12 months after the start of treatment.
Evaluation of reeptielization degree of the cervico-vaginal mucosa by a likert-type scale | 3,6 and 12 months
  A likert-type scale will be used to evaluate the reeptielization degree of the cervico-vaginal mucosa at 3, 6 and 12 months after the start of treatment.
Presence of HPV at 6 and 12 months after starting treatment. | 6 and 12 months]
  Percentage of patients with total and partial clearance of HPV measured by genotyping PCR at 6 and 12 months after starting treatment.
Evaluation of vaginal health status by vaginal health index score (Bachmann) | 3,6 and 12 months]
  The vaginal health index score (Bachmann) will be used to evaluate vaginal health status at 3, 6 and 12 months from the start of treatment
To evaluate the safety and tolerability of Papilocare® gel during the 6 months of treatment and 6 months of follow-up. | 6 and 12 months]
  Safety and tolerability: incidence, nature and severity of adverse events at 6 months of treatment and 6 months of follow-up period.
To assess the stress received from the patients at 3, 6 and 12 months after starting treatment. | 3,6 and 12 months]
  The stress will be assessed on the PSS14 scale (Perceived Stress Scale 14 items) at 3, 6 and 12 months after the starting treatment.
Evaluation of the satisfaction of papilocare gel use by a likert-type scale | 3 and 6 months]
  A likert-type scale will be used to evaluate the satisfaction of papilocare gel use by the patients at 3 and 6 months after the start of treat
Percentage of patients with good therapeutic compliance | 3 and 6 months]
  Percentage of patients with good adherence to the treatment will be used to evaluate the therapeutic compliance at 3 and 6 months after the start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Cortes Bordoy, MD, Study Chair — AEPCC
Locations (19):
- Spain (19):
  - Hospital U. de Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital Universitario HM Puerta del Sur, Móstoles, Madrid
  - Hospital Universitari Son Espases, Palma de Mallorca, Mallorca
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital General Universitario de Alicante, Alicante
  - Complejo Hospitalario Torrecárdenas, Almería
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d' Hebron, Barcelona
  - Hospital de Basurto, Bilbao
  - H. U. Reina Sofía, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Assir Hospitalet de Llobregat, L'Hospitalet de Llobregat
  - Hospital Universitario La Paz, Madrid
  - Hospital de Manacor, Manacor
  - H. R. U. de Málaga / Materno Infantil, Málaga
  - H. General Universitario Santa Lucía, Murcia
  - Hospital Virgen de la Macarena, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Álvaro Cunqueiro, Vigo

IPD SHARING:
Plan to Share IPD: Yes
The PIs from the participant sites gonna received the study protocol and the informed consent form previously to the initiation of the study and every time it occurs an amendment over the protocol, ICF or any other study document. Once the study has finished and the data has been analyzed, the PI's from the sites gonna received the CSR.
Supporting Information: Study Protocol, ICF, CSR